CLINICAL TRIAL: NCT05350813
Title: Impact of Procalcitonin-guided Algorithm on Early Discontinuation of Antibiotic Therapy in Pediatric Intensive Care Units : a Multicenter Randomized Controlled Trial
Brief Title: Impact of Procalcitonin-guided Algorithm on Early Discontinuation of Antibiotic Therapy
Acronym: PRODISCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/21/0334; 2022-A00246-37 (Other: ID-RCB)
Record Dates: First submitted 2022-04-15; First posted 2022-04-28 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Bacterial Infections
Keywords: procalcitonin; Children; Pediatric Intensive Care Unit; Procalcitonin-guided antibiotic therapy; Algorithm
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCT-guided arm (Experimental): Group of patients whose duration of antibiotic therapy will depend on procalcitonin (PCT) plasma levels on days 0 and 1, then on PCT plasma level every 48 hours and on patient clinical evolution evaluated by the fever, the infected organ, and the pSOFA (Pediatric Sequential Organ Failure Assessment) score every day until cessation of antibiotics in hospital or until discharge from hospital if the patient is discharged with an antibiotic treatment.
  Interventions: Procedure: Measurement of the PCT plasma levels
- standard-of-care arm (Active Comparator): A group of patients whose duration of antibiotic therapy will be determined by the type of infection, microbiological findings and clinical, biological and/or radiological course, according to standard practice based on guidelines.
  Interventions: Procedure: Usual practice based on guidelines

INTERVENTIONS:
Procedure: Measurement of the PCT plasma levels — antibiotic treatment duration will be based on PCT plasma levels
  Arms: PCT-guided arm
Procedure: Usual practice based on guidelines — antibiotic therapy duration will be determined by the type of infection, microbiological results and clinical, biological and/or radiological evolution, according to the usual practice based on guidelines.
  Arms: standard-of-care arm

SUMMARY:
In this randomized controlled open-label trial, conducted in 7 French Pediatric and Neonatal Intensive Care Units (ICUs), investigator team hypothesize that the use of a procalcitonin (PCT)-guided algorithm to discontinue antibiotic treatment will decrease antibiotic duration in critically ill children treated for a suspected or proven bacterial infection. Two hundred and ninety-six eligible patients will be randomly assigned in two groups: either PCT-guided or standard-of-care antibiotic discontinuation, and monitored over 28 days, until the end of their hospitalization, or up to the end of antibiotic treatment for bacterial infection recurrence occurring up to 28 days after the day of randomization.

DETAILED DESCRIPTION:
Infections are widespread in Pediatric and Neonatal ICU, and antibiotic treatments widely used. Long courses of antibiotic treatment increase the duration of hospitalization and are associated with changes in the microbiome, emergence of multidrug resistant organisms, and antibiotic-associated adverse events. In Pediatric and Neonatal ICU, PCT has a high negative predictive value to rule out bacterial infection. Thus, in sepsis patients and patients who initially appear to have sepsis but whose final diagnosis of bacterial infection is not retained, the use of a PCT-guided algorithm may be of value to shorten antibiotic duration without increasing infection recurrences. The algorithm has provided strong evidence of efficacy and safety among critically ill adults, excluding immunocompromised patients, patients with cystic fibrosis, and infections requiring prolonged antibiotic therapy. Similar data in critically ill children are lacking. A Spanish team from Sant Joan de Déu published three prospective non-randomized studies in Pediatric ICU (PICU), with encouraging results. Only one American randomized controlled trial (RCT) has been published in PICU with mixed results. One RCT is ongoing in India. Thus, our study will be the first French RCT to study the use of a PCT-guided algorithm to de-escalate antibiotic therapy in PICU, in order to provide evidence of efficacy and safety of such an algorithm in critically ill children with a suspected or proven bacterial infection. In addition, investigator team will also study the economic impact of a PCT-guided algorithm which has never been done before.

In the PCT-guided arm, PCT dosage will be done at Day 0 (day of randomization) and Day 1, and then every 48 hours until cessation of antibiotics in hospital or discharge from hospital if the patient is discharged with an antibiotic treatment. Antibiotic treatment will be stopped according to PCT value and patient clinical evolution. In the control group, antibiotic duration will be determined by usual practices based on guidelines. Inpatient evaluations will be conducted every day so long as patients receives antibiotics in hospital and usual clinical, biological and/or radiological monitoring will be conducted in both groups. To monitor infection recurrence occurring up to 28 days after the day of randomization and antibiotic-related adverse events, an evaluation will be conducted at the end of hospitalization, another at Day 28 (Day 0 = day of randomization), and a last at the end of antibiotic treatment bacterial infection recurrence, if the patient is discharged from hospital on or before Day 28 and is still treated with antibiotics for a bacterial infection recurrence at Day 28, or if the patient is discharged from hospital after Day 28 and is still treated for recurrence on the last day of hospitalization with antibiotics for a bacterial infection recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Neonates, infants and children hospitalized in Pediatric and Neonatal ICU and receiving intravenous antibiotics for less than 24 hours for an episode of suspected or proven community-acquired or nosocomial bacterial infection.
* Written informed consent signed by both parents or legal guardians.
* Affiliated to a social security scheme.
* Parents French-speaking.

Exclusion Criteria:

* Newborns <72 hours old.
* Neonates <37 weeks postmenstrual age.
* Age ≥18 years.
* Pregnant or breastfeeding women.
* Patients with cystic fibrosis.
* Immunocompromised patients including patients with hereditary immunodeficiency, agranulocytosis (neutrophils count <500/mm3), HIV infection with CD4 count <200/mm3, sickle cell disease, those who have undergone splenectomy, those who have a history of solid organ or hematopoietic stem cell transplant, those with hemopathy or solid organ tumor treated with chemotherapy, and those on immunosuppressive drugs including systemic corticosteroids taken daily for at least 15 days prior to Day 0.
* Inflammatory situations increasing PCT plasma concentrations in the absence of infection: burns, extracorporeal membrane oxygenation (ECMO), first 48 hours following an open-heart cardiac surgery with cardiopulmonary bypass.
* Infections requiring prolonged antibiotic therapy: infected thrombophlebitis, infective endocarditis, mediastinitis, abscess or empyema (e.g. peritonsillar abscess, retropharyngeal abscess, adenophlegmon, retroauricular abscess, retroorbital abscess, pulmonary abscess, pleural empyema, liver abscess, splenic abscess, brain abscess, subdural empyema, extradural empyema, epidural abscess, intramuscular abscess), necrotizing dermohypodermitis or necrotizing fasciitis, osteomyelitis, osteitis, arthritis, spondylodiscitis, prostatitis, tuberculosis, meningitis except those caused by Haemophilus and Meningococcus, infection on a device excluding intravascular catheter, endotracheal tube, tracheostomy, and urinary catheter.
* Antibiotic for prophylaxis.
* Children previously included in an interventional study in progress.

Ages: 3 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 296 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Total duration of antibiotic therapy (in days) for a suspected or proven bacterial infection, including the first episode and recurrences occurring within 28 days following the day of randomization | month 3 (maximum follow-up period of 3 months)
  Duration of antibiotic therapy (in days) including the length of treatment for recurrences occurring within 28 days following the day of randomization. The duration of antibiotic therapy for the first episode of suspected or proven bacterial infection is the time interval, expressed in days, between the starting time of intravenous antibiotics and the stopping time of the antibiotic therapy (intravenous, intramuscular or oral). The duration of antibiotic therapy for a recurrence of bacterial infection is the time interval, expressed in days, between the starting time of a new antimicrobial therapy (intravenous, intramuscular or oral) covering the initial causative bacteria within 28 days following the day of randomization, and the stopping time of this antibiotic therapy (even if ending after 28 days following the day of randomization).

SECONDARY OUTCOMES:
Total duration of broad-spectrum antibiotic therapy in days) for a suspected or proven bacterial infection, including the first episode and recurrences | month 3 (maximum follow-up period of 3 months)
  Duration of broad-spectrum antibiotic therapy (in days) including the length of treatment for recurrences occurring within 28 days following the day of randomization, and also the length of treatment for recurrences occurring within 28 days following the day of randomization. To identify broad-spectrum antibiotics, we used separately two definitions. Based on the historical definition, broad-spectrum antibiotics were all antibiotics except those with a useful activity against only Gram-positive bacteria (penicillin G, oxacillin, vancomycin, teicoplanin, linezolid, macrolides, clindamycin) and those whose main activity is against Gram-positive bacteria (amoxicillin, 1st generation cephalosporin [cefazolin, cephalexin], 2nd generation cephalosporin [cefuroxime, cefaclor, cefamandole], rifampicin).
Length of Intensive Care Unit stay (in days) from Day 0 (day of randomization) | month 3 (maximum follow-up period of 3 months)
  Length of Intensive Care Unit stay (in days) from Day 0 (day of randomization)
Length of hospital stay from Day 0 (day of randomization) | month 3 (maximum follow-up period of 3 months)
  Length of hospital stay from Day 0 (day of randomization)
Recurrence of bacterial infection within 28 days following the day of randomization | day 28
  Proportion of children with recurrence of bacterial infection within 28 days following the day of randomization. The recurrence of bacterial infection is defined as the isolation of one or more of the initial causative bacteria from the same or another site at 48 hours or more after cessation of antibiotics, combined with clinical signs or symptoms of infection, or the need to prescribe a new antimicrobial therapy covering this pathogen. All recurrences of bacterial infection occurring up to Day 28, and treated in hospital (same hospital stay as for the first episode, or new hospital stay) or in ambulatory care, will be taken into account.
All cause mortality at Day 28 (Day 0 = day of randomization) | day 28
  All cause mortality rate at Day 28 (Day 0 = day of randomization). All-cause mortality is a measure of all deaths, due to any cause, that occur during a clinical study.
All cause mortality at the end of antibiotic treatment for bacterial infection recurrence (if ending after Day 28) | month 3 (maximum follow-up period of 3 months)
  All cause mortality rate at the end of antibiotic treatment for bacterial infection recurrence (if ending after Day 28). All-cause mortality is a measure of all deaths, due to any cause, that occur during a clinical study.
Sepsis-related mortality at Day 28 (Day 0 = day of randomization) | day 28
  Sepsis-related mortality rate at Day 28 (Day 0 = day of randomization). Sepsis-related mortality is a measure of all deaths related to the first bacterial infection episode or bacterial infection recurrence, that occur during the study.
Sepsis-related mortality at the end of antibiotic treatment for bacterial infection recurrence (if ending after Day 28). | month 3 (maximum follow-up period of 3 months)
  Sepsis-related mortality rate at the end of antibiotic treatment for bacterial infection recurrence (if ending after Day 28). Sepsis-related mortality is a measure of all deaths related to the first bacterial infection episode or bacterial infection recurrence, that occur during the study.
Antibiotic-related adverse events | month 3 (maximum follow-up period of 3 months)
  Antibiotic-related adverse events
Adherence to the PCT-guided algorithm | month 3 (maximum follow-up period of 3 months)
  This outcome will be evaluated by a stop of antibiotics within 24 hours after reaching stopping criteria : - Before Day 3: PCT levels at Day 0 and Day 1 less than 0.5 ng/mL.; - Starting Day 3: PCT level less than 0.5 ng/mL or down by ≥80% from the peak value since Day 0 AND favorable patient clinical course (defined by a decrease in pSOFA score compared to maximal value at Day 0 or Day 1, a reduction of fever and an improvement of the infected organ). - Or if the antibiotic duration, as defined by current infectious guidelines, is reached and the patient shows a favorable course, even if PCT is still ≥0.5 ng/mL or >20% of the peak value.
Incremental cost-effectiveness ratios | month 3
  This outcome will be expressed in terms of hospital costs per number of patients without recurrent bacterial infection at 3 months and hospital costs per number of patients alive at 3 months
Costs of antibiotic therapy and PCT testing during each inpatient stay | month 3
  Costs of antibiotic therapy and PCT testing during each inpatient stay

CONTACTS AND LOCATIONS:
Overall Officials: Romain AMADIEU, MD, Principal Investigator — University Hospital of Toulouse
Locations (7):
- France (7):
  - CHU Amiens Picardie, Amiens
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de NANTES, Nantes
  - APHP, Paris
  - CHU La Réunion, Saint-Denis
  - University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No